CLINICAL TRIAL: NCT03272490
Title: Polyaxial Locking Plates in Treating Distal Humeral Fractures: a Comparative Randomized Trial for Clinical Outcome
Brief Title: Polyaxial Locking Plates in Treating Distal Humeral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Chlodwig Kirchhoff, Principal Investigator, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Distal Humerus Fracture
Keywords: locking plate; anatomical preshaped; polyaxial; outcome
MeSH Terms: conditions — Humeral Fractures, Distal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medartis (Active Comparator): Surgery using the Medartis Implant
  Interventions: Procedure: Medartis
- Synthes (Active Comparator): Surgery using the Synthes implant
  Interventions: Procedure: Synthes

INTERVENTIONS:
Procedure: Medartis — Surgery using the medartis implant
  Arms: Medartis
Procedure: Synthes — Surgery using the Synthes implant
  Arms: Synthes

SUMMARY:
20 patients with distal humeral fractures (AO 13-A1 - AO 13-C3) were included in the current study since 2014. After completing the randomization plan, patients were distributed into two groups for different variable angle locking plates (DePuy Synthes VA-LCP vs. Medartis Aptus Elbow). Clinical and radiological follow-ups were conducted 6 weeks, 12 weeks, 6 months and 12 months after the operation.

DETAILED DESCRIPTION:
Before study initiation the approval of the local ethics committee of (Trial Number 253/14) was obtained. The clinical trial included 20 patients with fractures of the distal humerus recruited from a level-one university trauma centre. Patient recruitment was conducted between 03/2014 and 12/2015. Fractures of the distal humerus, as defined by the AO classification system (AO 13-A1 - AO 13-C3), were included in this study as they were identified by the treating surgeon being applicable for locking plate treatment and after written informed consent of the patients was obtained. All patients were randomized following a randomization plan (Randlist, DatInf GmbH, Tübingen, Germany) for either being treated with the DePuy Synthes VA-LCP 2.7/3.5 mm (DePuy Synthes, Umkirch, Germany) or with the Medartis Aptus Elbow system 2.0/3.8 mm (Medartis, Basel, Switzerland). Both systems include anatomically preshaped, polyaxial angular stable locking plates in various sizes. Angle stable screw positioning with the freedom of +/- 15° off-axis screw placement gives the surgeon a large variety in both systems.

The inclusion criteria involve all patients from the age of 18 to 95 years who suffered from a distal humeral fracture (AO 13-A1 - AO 13-C3) that had to undergo operative treatment. The exclusion criteria involve all under-aged patients (< 18 years), pregnant patients and patients with a mental disorder as well as patients under comprehensive legal support. In addition, pathological fractures had been excluded from the study.

Surgical technique

All patients were operated by experienced upper extremity surgeons. The mean interval between injury and operation was 2.4 days (range 0-12 days). General anaesthesia was used in all cases and a single dose of 1.5 mg cephalosporin was given preoperatively for prophylaxis. Patients were positioned in prone position with the injured arm on a radiolucent, small padded arm holder. Under tourniquet control, the posterior approach (Bryan-Morrey) to the distal humerus was performed in all cases. Additional olecranon osteotomy was performed in 7 cases (3x DePuy Synthes vs. 4x Medartis Aptus Elbow) presenting with AO type 13 C2 and AO type 13 C3 fractures. Postoperatively, physiotherapy was initiated using the same rehabilitation protocol for both groups. Passive and active assisted ROM was permitted immediately without limitations, while weight bearing was restricted for 6 weeks.

Follow-up evaluation

All patients were initially followed-up 6 weeks after operation. Additional follow-ups were performed 3, 6 and 12 months postoperatively. The follow-up examinations were carried out by an independent investigator not involved in patient´s initial surgical treatment (MC). After the assessment of pain using the visual analogue scale (VAS) was documented, ROM and collateral ligament stability were documented on standardized scoring sheets. For subjective evaluation, patients rated their satisfaction for elbow use on a scale of 1 to 6 (1-highly satisfied; 2-satisfied; 3-moderate; 4-sufficient; 5-unsatisfied; 6-very unsatisfied). Moreover, sensomotoric disturbances and postoperative complications were recorded. For functional upper extremity and elbow scoring the shortened Disabilities of the Arm, Shoulder and Hand Score (QuickDASH) and the Mayo Elbow Performance Score (MEPS) were comprised. Postoperative x-rays were evaluated with special respect to bony healing, secondary loss of reduction and heterotopic ossifications.

Statistics

Statistical analyses were performed using the statistical software SigmaStat (version 3.5; Systat Software, San Jose, CA, USA). The scores at certain time points were compared with an independent t test after a normality check had been passed and equal variances had been detected. Normal distributed data with unequal variances would have been compared with Welch's t test. Arbitrarily data was tested with Mann-Whitney U test. The significance level was set at p= 0.05.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria involve all patients from the age of 18 to 95 years who suffered from a distal humeral fracture (AO 13-A1 - AO 13-C3) that had to undergo operative treatment

Exclusion Criteria:

* The exclusion criteria involve all under-aged patients (< 18 years), pregnant patients and patients with a mental disorder as well as patients under comprehensive legal support. In addition, pathological fractures had been excluded from the study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Mayo Elbow Performance Score (MEPS) | 12 months
  clinical and functional outcome

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bibethaler, Prof., Study Director — Department of Trauma Surgery Klinikum rechts der Isar Technical University of Munich, Germany Ismaninger Strasse 22 81675 Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cronlein M, Lucke M, Beirer M, Pforringer D, Kirchhoff C, Biberthaler P, Braun KF, Siebenlist S. Polyaxial locking plates in treating distal humeral fractures: a comparative randomized trial for clinical outcome. BMC Musculoskelet Disord. 2017 Dec 28;18(1):547. doi: 10.1186/s12891-017-1910-9. PMID 29282027